CLINICAL TRIAL: NCT06996691
Title: A Comparative Study of Erector Spinae Plane Block Versus Serratus Anterior Plane Block for Postoperative Analgesia After Video-assisted Thoracoscopic Surgery
Brief Title: Erector Spinae Plane Block Versus Serratus Anterior Plane Block in VATS
Acronym: VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 145/2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: Video Assisted Thoracic Surgery (VATS)
Keywords: VATS; Erector spinae plane block; Serratus anterior plane block
MeSH Terms: interventions — Population Groups; Saposins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Erector spinae block group (Active Comparator): After selecting the target transverse process for the nerve block, place the transducer in a paramedian sagittal orientation, approximately 2cm away from the midline (spinous processes), and try to vizualize the transverse process at the level of T5 Complete the nerve block with 30ml of 0.25% levobupivacaine for erector spinae block
  Interventions: Procedure: Erector Spinae Plane Block (ESPB) group
- group B: Serratus anterior block group (Active Comparator): High-frequency linear transducer should be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib. With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized.
  Then, using ultrasound guidance, the needle is advanced in-plane and the local anesthetic is injected anteriorly to the rib and deep to the serratus anterior.
  After opening the fascial plane, a volume of dilute local anesthetic, 30 mL of 0.25% levobupivacaine, should be gradually injected.
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB) group

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESPB) group — 30ml of 0.25% levobupivacaine for erector spinae block at level of T5
  Arms: Group A: Erector spinae block group
Procedure: Serratus Anterior Plane Block (SAPB) group — 30 mL of 0.25% levobupivacaine injected anteriorly to the rib and deep to the serratus anterior at level of 5 th rib
  Arms: group B: Serratus anterior block group

SUMMARY:
Pain control remains challenging in patients undergoing video-assisted thoracoscopic surgery (VATS). It is advised to use a regional block to lower postoperative opioid usage. This study evaluates efficacy of Erector spinae plane (ESP) block in comparison to Serratus anterior plane block (SAP) in pain management for patients undergoing video-assisted thoracoscopic surgery(VATS).

DETAILED DESCRIPTION:
Minimally invasive thoracic surgery (MITS) has become more common over the past decade, with the proportion of lung resections performed using this technique increasing from 16% in 2005 to 47% in 2015.

VATS is a minimally invasive procedure that allows rapid recovery compared to thoracic surgery. Patients scheduled for VATS experience moderate to severe pain following the procedure. This represents a significant burden peri-operatively as there is a strong relationship between poor pain control and the development of complications like pneumonia and atelectasis due to interference with spontaneous deep breathing & coughing. These complications have a negative impact on functional recovery; therefore, adequate postoperative pain relief assists in improving functional outcomes & accelerates hospital discharge.

Multimodal techniques for pain control have been recommended by The American Society of Anesthesiologists (ASA) for the management of acute postoperative pain. Traditional analgesia based on opioids have multiple adverse effects such as respiratory depression, nausea, vomiting, itching and dizziness.

SAP block was first described in 2013 by Blanco as an analgesic technique.it is proposed to block the lateral cutaneous branch of the intercostal nerve, long thoracic nerve, and dorsal thoracic nerve. The block range of the SAPB covers the incisions of video-assisted thoracoscopic surgery (VATS) and the site of the chest tube, which are often located in the antero-lateral chest wall. The local anaesthetic injection was described in two planes: the 'superficial plane' and deep plane.

An ultrasound-guided ESP block was firstly reported in 2016. The ESP block injects a local anaesthetic around the erector spinae muscle at approximately the level of the T5. It may be able to block the dorsal and ventral rami of the thoracic spinal nerves. The first report of the successful use of this procedure was in 2016; the block was used to manage thoracic neuropathic pain in a patient with metastatic disease of the ribs and rib fractures

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI)=18 to 40 kg/m2

Exclusion Criteria:

* Contraindications to regional anesthesia as bleeding disorders , allergy to local anesthetic or infection at block site
* pre-existing chronic pain
* history of opiate abuse
* sepsis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
post operative opioid consumption | 24 hours post operative
  post operative meperidine consumption throughout

SECONDARY OUTCOMES:
intraoperative fentanyl consumption | during the surgery
  total introperative fentanyl dose
the numerical rating scale | 24 hours post operative
  a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 to 10 integers) that best reflects the intensity of their pain. 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable")

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF